CLINICAL TRIAL: NCT04476836
Title: Animal-Assisted Therapy in Middle-aged and Older Patients With Schizophrenia
Brief Title: Animal-Assisted Therapy in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202000549B0
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia; Animal-assisted Therapy
Keywords: schizophrenia; animal-assisted therapy
MeSH Terms: conditions — Schizophrenia | interventions — Animal Assisted Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAT group (Experimental): Animal-assisted therapy will be provided one 1-hour session per week for 48 weeks.
  Interventions: Other: Animal-Assisted Therapy
- control group (No Intervention): routine care

INTERVENTIONS:
Other: Animal-Assisted Therapy — Animal-Assisted Therapy is when animals are used in goal-directed treatment sessions. These goals can be physical, mental, emotional or social.
  Arms: AAT group

SUMMARY:
Animal-assisted therapy (AAT) can be helpful to improve the psychiatric, emotional, physical,and social status in patients with physical and mental illness and the elderly.

The study aims to investigate the effects of AAT program in middle-aged and older patients with schizophrenia. The investigators will recruit 40 patients with schizophrenia in psychiatric ward randomised into AAT group and control group. AAT group will complete the 12-week program. This study contains two assessment sessions before and after intervention, including PANSS, ACIS, MoCA-T, CHI, DASS-21, CST, TUG and 5MWT.

DETAILED DESCRIPTION:
Animal-assisted therapy (AAT) can be helpful to improve the outcomes of psychiatric and emotional symptoms, physical activeness, social skills, well-beings in patients with physical and mental illness and the elderly.

The study aims to assess the applications and outcomes of psychiatric symptoms, social skills, cognitive function, well-beings, emotional status and physical fitness of AAT program applied to middle-aged and older patients with chronic schizophrenia.

The investigators will recruit 40 patients with chronic schizophrenia who were admitted to day care ward and rehabilitation ward, and conduct a randomized, controlled study. 40 patients will be stratified by the ward into AAT group and control group. AAT group will complete the 12-week program. This study contains two assessment sessions completed within one week before and after 12-week program. Subjects will be evaluated by the PANSS, ACIS, MoCA-T, CHI, DASS-21, CST, TUG and 5MWT in both sessions. Statistical analysis is examined using paired t-test to see whether there is a significant difference (based on p-value) between the scores of two assessment sessions in the AAT and control group, and using independent t-test to see whether there is a significant difference in the change scores of two assessment sessions between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of schizophrenia according to the DSM-5.
2. Adult aged 40 years or older.
3. Having stable physical and psychological health conditions based on master clinician judgment.
4. Having the will to participate in the study after thorough comprehension of the content.
5. Not receiving treatment protocol last half a year.

Exclusion Criteria:

1. Severe cognitive impairment e.g. aphasia, being unable to follow 3 or more orders.
2. Being allergic to animals.
3. History of Asthma.
4. Coagulation disorders
5. presenting symptoms of specific phobia, anxiety disorder and obsessive-compulsive disorder in context of dog, infection and contamination.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-08-24 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change scores of Positive and Negative Syndrome Scale | Baseline, immediate after treatment
  This test is used for measuring symptom severity of patients with schizophrenia.

SECONDARY OUTCOMES:
Change scores of The Assessment of Communication and Interaction Skills | Baseline, immediate after treatment
  This test is an observational rating scale designed to measure communication and interaction skills.
Change scores of The Taiwanese version of Montreal Cognitive Assessment | Baseline, immediate after treatment
  This test is a cognitive screening test in the detection of mild cognitive impairment and Alzheimer's disease.
Change scores of Chinese Happiness Inventory | Baseline, immediate after treatment
  This test is a subjective measure of well-being.
Change scores of Depression Anxiety Stress Scales-21 | Baseline, immediate after treatment
  This test is a 21-item self report instrument for measuring depression, anxiety and tension/stress.
Change scores of Chair Stand Test | Baseline, immediate after treatment
  This test is to measure leg strength.
Change scores of Timed Up and Go | Baseline, immediate after treatment
  This test is to assess mobility, balance, walking ability, and fall risk in older adults.
Change scores of The 5-Meter Walk Test | Baseline, immediate after treatment
  This test is to assess walking speed.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung Medical Center, Kaohsiung City, Taiwan